CLINICAL TRIAL: NCT00785512
Title: A Prospective, Randomized, Double-Blind, Placebo Controlled Study of the Long-Term Efficacy of Nebivolol in Hypertensive Patients After Withdrawal of Therapy
Brief Title: A Study on the Long-term Efficacy of Nebivolol After Withdrawal of Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: John Whalen, MD, Executive Director, Clinical Development, Cardiovascular, Forest Research Institute, a subsidiary of Forest Laboratories Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEB-MD-17
Record Dates: First submitted 2008-11-03; First posted 2008-11-05 (Estimated); Results first posted 2010-09-15 (Estimated); Last update posted 2010-09-15 (Estimated); Status verified 2010-08

CONDITIONS: Hypertension
Keywords: nebivolol; Bystolic®; Hypertension; blood pressure; withdrawal
MeSH Terms: conditions — Hypertension | interventions — Nebivolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Nebivolol 10 mg, 10-mg Nebivolol nontrade tablets , oral administration Nebivolol 20 mg, 20-mg Nebivolol nontrade tablets , oral administration Nebivolol 40 mg, two 20-mg Nebivolol nontrade tablets , oral administration
  Interventions: Drug: Nebivolol
- 2 (Placebo Comparator): Matching placebo tablets, oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nebivolol — Nebivolol 10 mg, 10-mg Nebivolol nontrade tablets , oral administration Nebivolol 20 mg, 20-mg Nebivolol nontrade tablets , oral administration Nebivolol 40 mg, two 20-mg Nebivolol nontrade tablets , oral administration
  Other Names: Bystolic® (nebivolol)
  Arms: 1
Drug: Placebo — Matching placebo tablets, oral administration
  Arms: 2

SUMMARY:
This study will evaluate the long-term efficacy of nebivolol monotherapy in patients with stage 1 or stage 2 hypertension after the withdrawal of active medication.

ELIGIBILITY:
Inclusion Criteria:

* male and female outpatients 18 to 79 years of age
* Females must be post-menopausal, or not pregnant and using an approved contraceptive regimen
* meet criteria for stage I or II hypertension
* currently not treated, or being treated with no more than two anti-hypertensive medications

Exclusion Criteria:

* type 1 or type 2 diabetes
* secondary hypertension
* evidence of other concurrent disease or conditions that might interfere with the conduct of the study
* treatment with any investigational study drug within 30 days of Screening (Visit 1)
* have a history of hypersensitivity to nebivolol or other β-blockers

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2008-11; Primary Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tatjana Lukic, MD, MSc, Study Director — Forest Research Institute, a Subsidiary of Forest Laboratories Inc.
Locations (23):
- United States (23):
  - Forest Investigative Site, Chandler, Arizona
  - Forest Investigative Site, Phoenix, Arizona
  - Forest Investigative Site, Los Angeles, California
  - Forest Investigative Site, Bradenton, Florida
  - Forest Investigative Site, Brooksville, Florida
  - Forest Investigative Site, DeLand, Florida
  - Forest Investigative Site, Hollywood, Florida
  - Forest Investigative Site, Miami, Florida
  - Forest Investigative Site, Pembroke Pines, Florida
  - Forest Investigative Site, St. Petersburg, Florida
  - Forest Investigative Site, Auburn, Maine
  - Forest Investigative Site, Cary, North Carolina
  - Forest Investigative Site, Hickory, North Carolina
  - Forest Investigative Site, Salisbury, North Carolina
  - Forest Investigative Site, Wilmington, North Carolina
  - Forest Investigative Site, Winston-Salem, North Carolina
  - Forest Investigative Site, Cincinnati, Ohio
  - Forest Investigative Site, Marion, Ohio
  - Forest Investigative Site, Lancaster, Pennsylvania
  - Forest Investigative Site, Mt. Pleasant, South Carolina
  - Forest Investigative Site, Simpsonville, South Carolina
  - Forest Investigative Site, New Tazewell, Tennessee
  - Forest Investigative Site, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was five months, from November 2008 through March 2009.
Pre-assignment Details: Patients went through a 4-5 week, single blind, placebo run-in/washout phase, followed by a 12 week single-blind active treatment phase with nebivolol before randomization
Period: Overall Study
Arm/Group | Nebivolol | Placebo
Started | 102 | 105
Completed | 99 | 101
Not Completed | 3 | 4
Not completed — Inclusion/Exclusion not meet | 0 | 0
Not completed — Adverse Event | 0 | 0
Not completed — Lack of Efficacy | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 3 | 0
Not completed — Precedure Refused | 0 | 0
Not completed — IVRS Programing Error | 0 | 0
Not completed — Physician Decision | 0 | 0
Not completed — Lack of compliance | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nebivolol | Placebo | Total
Number analyzed (Participants) | 102 | 105 | 207
Age Categorical [Number; unit: participants]
  <18 years | 0 | 0 | 0
  Ages 18 to 64 years | 86 | 91 | 177
  >=65 years | 16 | 14 | 30
Age Continuous [Mean (Standard Deviation); unit: years] | 52.6 (11.2) | 52.9 (10.2) | 52.8 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 43 | 86
  Male | 59 | 62 | 121
Region of Enrollment [Number; unit: participants]
  United States | 102 | 105 | 207

OUTCOME MEASURES:

1. Primary Outcome: Trough Sitting Diastolic Blood Pressure
Description: Change from baseline, week 0 (Visit 9) to Week 4 (Visit 12) in peripheral diastolic blood pressure measured at drug trough.
Time Frame: From baseline, week 0 (Visit 9) to week 4 (Visit 12)
Measure: Mean (Standard Deviation); unit: mm HG
Arm/Group | Nebivolol | Placebo
Number analyzed (Participants) | 101 | 105
mm HG
  Baseline | 81.3 (7.2) | 81.1 (7.0)
  Change from baseline | 1.8 (7.3) | 7.7 (8.6)

2. Secondary Outcome: Trough Sitting Systolic Blood Pressure
Description: Change from baseline, week 0 (Visit 9) to Week 4 (Visit 12) in peripheral systolic blood pressure measured at drug trough.
Time Frame: From baseline, week 0 (Visit 9) to week 4 (Visit 12)
Measure: Mean (Standard Deviation); unit: mm HG
Arm/Group | Nebivolol | Placebo
Number analyzed (Participants) | 101 | 105
mm HG
  Baseline | 134.1 (12.5) | 134.4 (11.4)
  Change from baseline | 3.5 (12.3) | 7.6 (11.8)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for a period of 9 months, from November 2008 to August 2009.
Groups:
- Single-blind Nebivolol: Pre-randomization 12 week nebivolol treatment.
Arm/Group | Single-blind Nebivolol | Nebivolol | Placebo
Serious Adverse Events (participants affected / at risk) | 2/269 | 0/102 | 0/105
Other Adverse Events (participants affected / at risk) | 29/269 | 0/102 | 0/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single-blind Nebivolol (N=269) | Nebivolol (N=102) | Placebo (N=105)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single-blind Nebivolol (N=269) | Nebivolol (N=102) | Placebo (N=105)
Bradycardia (Cardiac disorders) | 16 | 0 | 0
Nasopharyngitis (Infections and infestations) | 14 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor can review results communications prior to public release & can embargo communications re: results for 60 days from time submitted to sponsor for review. PI shall not disclose sponsor's confidential information. Upon sponsor's request, PI shall delete any proprietary info & shall not include raw data in the publication. On sponsor's request, PI shall delay submission for any pub while sponsor files patent applications. Any publication will give recognition to Sponsor's support.